CLINICAL TRIAL: NCT04663698
Title: Evaluation of PLB Physiology in COPD - Untersuchung Zur Physiologie Der Lippenbremse Bei COPD
Brief Title: The Effect of Volitional Pursed-lips Breathing
Acronym: PLB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karl Josef Franke, PD DR med (Industry)
Responsible Party: Sponsor-Investigator, Karl Josef Franke, PD DR med, Clinical Director, Institut für Pneumologie Hagen Ambrock eV
Organization: Institut für Pneumologie Hagen Ambrock eV (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PLB2019
Record Dates: First submitted 2020-10-22; First posted 2020-12-11 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: COPD
Keywords: Pursed-lips Breathing; Resistor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy (Experimental): Lung-healthy subjects, randomized lung function testing
  Interventions: Other: Baseline; Other: MESH-Resistor 5; Other: MESH-Resistor 10; Other: Perforated Resistor 7; Other: Perforated Resistor 11
- Patient 1 (Experimental): COPD patients, randomized lung function testing
  Interventions: Other: Baseline; Other: MESH-Resistor 5; Other: MESH-Resistor 10
- Patient 2 (Experimental): COPD patients, randomized lung function testing
  Interventions: Other: Baseline; Other: Perforated Resistor 7; Other: Perforated Resistor 11
- Patient 3 (Experimental): COPD patients, randomized lung function testing
  Interventions: Other: Baseline; Other: MESH-Resistor 5; Other: Perforated Resistor 7
- Patient 4 (Experimental): COPD patients, randomized lung function testing
  Interventions: Other: Baseline; Other: MESH-Resistor 5; Other: Perforated Resistor 11

INTERVENTIONS:
Other: Baseline — Lung function testing with MasterScreen™ Body, CareFusion Germany GmbH
Other: MESH-Resistor 5 — Lung funtion testing with MasterScreen™ Body, CareFusion Germany GmbH, Mouthpiece with mesh-resistor (5hPa/L) to create laminar airflow
  Other Names: Rudolph Flow Resistance Standards; HANS RUDOLPH, Inc.
  Arms: Healthy; Patient 1; Patient 3; Patient 4
Other: MESH-Resistor 10 — Lung funtion testing with MasterScreen™ Body, CareFusion Germany GmbH, Mouthpiece with mesh-resistor (10hPa/L) to create laminar airflow
  Other Names: Rudolph Flow Resistance Standards; HANS RUDOLPH, inc
  Arms: Healthy; Patient 1
Other: Perforated Resistor 7 — Lung function testing with MasterScreen™ Body, CareFusion Germany GmbH, Mouthpiece with perforated resistor (inside diameter 7mm) to create a turbulent airflow
  Other Names: 900MR405; Fisher&Paykel Healthcare
  Arms: Healthy; Patient 2; Patient 3
Other: Perforated Resistor 11 — Lung function testing with MasterScreen™ Body, CareFusion Germany GmbH, Mouthpiece with perforated resistor (inside diameter 11mm) to create a turbulent airflow
  Other Names: 900MR406; Fisher&Paykel Healthcare
  Arms: Healthy; Patient 2; Patient 4

SUMMARY:
Simulation of pursed-lips breathing by defined stenoses in pulmonary function diagnostics to quantify the effect of the pursed-lips breathing

DETAILED DESCRIPTION:
Since many years it is recommended for COPD patients to reduce the crossdiameter of the lips in order to improve the exhalation by means of so-called pursed-lips breathing (PLB). But the effects have never been studied quantitatively. In this study, the PLB effect is simulated during lung function diagnostics, using different sized resistors inserted into the routine mouthpiece of the flow sensor to resemble the effective airway resistances of a PLB maneuver. This prospective, randomized study includes 20 healthy subjects and 50 COPD patients, who will perform lung function testing with 4 different sized resistors.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* COPD (GOLD I- IV)
* Stable respiratory situation that allows routine lung funtion
* capable of communication

Healthy:

* Lung Healthy
* capable of communication

Exclusion Criteria:

* Invasive Ventilation
* Other serious acute physical illnesses that require immediate intensive medical treatment
* Acute hypercapnic decompensation with a pH < 7.35 in the capillary BGA
* Pregnancy or Nursing
* Not able to give consent
* Not willing or able to follow the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Lung function parameter FEV1 | up to 1 hour
  Measuring of lung function parameters with different resistors to simulate PLB unit: L, measured with der MasterScreen™ Body, CareFusion

SECONDARY OUTCOMES:
PEF - expiratory Peak Flow | up to 1 hour
  unit: L, measured with der MasterScreen™ Body, CareFusion
RV%TLC | up to 1 hour
  unit: %, measured with der MasterScreen™ Body, CareFusion

CONTACTS AND LOCATIONS:
Locations (1):
- Märkische Kliniken GmbH, Klinikum Lüdenscheid, Lüdenscheid, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No